CLINICAL TRIAL: NCT04350606
Title: A MULTICENTER, OPEN-LABEL, SINGLE-ARM STUDY TO ASSESS THE EFFICACY AND SAFETY OF PF-06462700 ADMINISTERED INTRAVENOUSLY AT 40 MG/KG/DAY FOR 4 DAYS IN JAPANESE PARTICIPANTS WITH MODERATE AND ABOVE APLASTIC ANEMIA
Brief Title: A Study to Assess Efficacy and Safety of PF-06462700 in Japanese Participants With Aplastic Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B5411003; ATGAM Japan local ph3 study (Other: Alias Study Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-17 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia, globulin, ATG, Anti-human Thymocyte Immunogloblin
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-006462700 group (Experimental): All enrolled participants will be administrated PF-006462700.
  Interventions: Biological: PF-06462700

INTERVENTIONS:
Biological: PF-06462700 — PF-06462700 is classified as an immunosuppressant/ immunosuppressive agent. It is the purified, concentrated, and sterile gamma globulin, primarily monomeric immunoglobulin G (IgG), from hyperimmune serum of horses that are immunized with human thymus lymphocytes.
  Other Names: Brand name in the US: ATGAM

SUMMARY:
The purpose of the study is to assess the efficacy and safety of PF-06462700 administered intravenously at 40 mg/kg/day for 4 days in Japanese participants with moderate and above aplastic anemia for making an approval application in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 2 years and more, inclusive, at Visit

  1 (Screening).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Have a clinical diagnosis of aplastic anemia by bone marrow aspiration/biopsy findings and/or magnetic resonance imaging (MRI) etc.
* Must meet the following criteria of moderate and above aplastic anemia
* Capable of giving signed informed consent/assent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD)/assent document and in this protocol.

Exclusion Criteria:

* Eligible and willing to have a sibling allogeneic stem cell transplantation.
* Evidence of a myelodysplastic syndrome (except for refractory cytopenia in children), as well as other primitive marrow disease.
* History or clinical suspicion of congenital aplastic anemia (Fanconi anemia, Congenital keratosis, etc).
* History of malignant tumors with active disease within 5 years from study participation.
* Participants who are clearly infected with hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), and human T-cell leukemia virus type

  1 (HTLV-1).
* Pregnant or breast-feeding participants.
* Participants with severe hepatic, renal or cardiac failure, or any other life-threatening concurrent [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or total bilirubin values >5 × upper limit of normal (ULN), and/or creatinine value >2 × ULN].
* Participants with hypersensitivity such as shock after skin test of this study drug.
* Participants with uncontrolled severe infection (pneumonia, sepsis, etc).
* Participants who received live vaccine or live attenuated vaccine within 6 weeks prior to the first dose of study drug.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Prior immunosuppressive therapy with lymphocyte-depleting agents/therapies, including both non-B-cell selective and B-cell-depleting agents (e.g., alefacept, alemtuzumab, rituximab). However, participants previously treated with rATG may enroll.
* Previous history of stem cell transplantation.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
* Baseline 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (e.g., baseline corrected QT [QTc] interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Keio University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kanda Y, Mori T, Narita A, Wolter KD, Yoshimatsu H, Nishimura K. Efficacy and safety of equine anti-thymocyte immunoglobulin (eATG) in three Japanese patients with moderate to very severe aplastic anemia: a case series. Int J Hematol. 2023 Jan;117(1):37-43. doi: 10.1007/s12185-022-03496-5. Epub 2022 Nov 28. PMID 36441357
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5411003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 3 participants signed the inform consent form (ICF). Out of which 0 participants were screen failures, 3 actually enrolled into the study and assigned to a study treatment.
Groups:
- PF-06462700: Participants aged 2 years or greater than (>) 2 years with moderate and above severity aplastic anemia received PF-06462700 at a dose of 40 milligram per kilogram per day (mg/kg/day), intravenously (IV) for 4 days. Participants after treatment were followed up for 24 weeks.
Period: Overall Study
Arm/Group | PF-06462700
Started | 3
Treated | 3
Follow-up | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants assigned to investigational product and who took at least 1 dose of investigational product.
Groups:
- PF-06462700: Participants aged 2 years or >2 years with moderate and above severity aplastic anemia received PF-06462700 at a dose of 40 mg/kg/day, IV for 4 days. Participants after treatment were followed up for 24 weeks.
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.67 (16.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematologic Response at Week 12
Description: Hematologic response was considered to be "effective" when 2 or more of the following criteria were met: absolute neutrophil count greater than or equal to (>=) 500 per microliters, platelet count >=20,000 per microliters and reticulocyte count >=60,000 per microliters was observed. In this outcome measure, number of participants with hematologic response classified as effective and not effective were reported. Improvement in counts that were dependent upon exogenously administered growth factors or transfusion, was not considered as fulfilling response criteria.
Time Frame: Week 12 Follow-up Visit
Population: Full analysis set (FAS) included participants were assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Participants
  Effective | 2
  Not Effective | 1

2. Secondary Outcome: Number of Participants With Hematologic Response at Week 24
Description: Hematologic response was considered to be "effective" when 2 or more of the following criteria were met: absolute neutrophil count >=500 per microliters, platelet count >=20,000 per microliters and reticulocyte count >=60,000 per microliters was observed. In this outcome measure, number of participants with hematologic response classified as effective and not effective were reported. Improvement in counts that were dependent upon exogenously administered growth factors or transfusion, was not been considered as fulfilling response criteria.
Time Frame: Week 24 Follow-up Visit
Population: FAS included participants who were assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Participants
  Effective | 2
  Not Effective | 1

3. Secondary Outcome: Absolute Neutrophil Count at Day 4, Weeks 1, 2, 4, 6, 8, 10, 12, 24
Time Frame: Treatment: Day 4; Follow-up: Week 1, 2, 4, 6, 8, 10, 12, 24
Population: as for outcome 2
Measure: Number; unit: Neutrophil cells per microliter
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Neutrophil cells per microliter | NA — It was planned data would not be summarized. Individual data cannot be reported for this outcome measure because they are directly personal information.

4. Secondary Outcome: Platelet Count at Day 4, Weeks 1, 2, 4, 6, 8, 10, 12, 24
Time Frame: Treatment: Day 4; Follow-up: Week 1, 2, 4, 6, 8, 10, 12, 24
Population: as for outcome 2
Measure: Number; unit: Platelet cells per microliter
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Platelet cells per microliter | NA — It was planned data would not be summarized. Individual data cannot be reported for this outcome measure because they are directly personal information.

5. Secondary Outcome: Reticulocyte Count at Day 4, Weeks 1, 2, 4, 6, 8, 10, 12, 24
Time Frame: Treatment: Day 4; Follow-up: Week 1, 2, 4, 6, 8, 10, 12, 24
Population: as for outcome 2
Measure: Number; unit: Reticulocyte cells per microliter
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Reticulocyte cells per microliter | NA — It was planned data would not be summarized. Individual data cannot be reported for this outcome measure because they are directly personal information.

6. Secondary Outcome: Number of Participants Who Survived During the Study
Description: In this outcome measure, number of participants who survived during the study were observed.
Time Frame: Screening (up to 28 days prior to Day 1 of treatment) up to 24 weeks of follow-up (approximately up to 28 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Participants | 3

7. Secondary Outcome: Number of Participants With Transfusion Independence at Weeks 12 and 24
Description: Transfusion independence at Week 12 was defined as when participants did not have any transfusion records from the time of the first dose of the investigational product at Day 1 to the day of Week 12 follow-up visit (inclusive). Transfusion independence at Week 24 was defined as when participants did not have any transfusion records from the day after Week 12 follow-up visit to the day of Week 24 follow-up visit (inclusive).
Time Frame: Week 12 Transfusion Independence: Day 1 of Treatment up to Week 12 Follow-up Visit (approximately 12 weeks); Week 24 Transfusion Independence: Day after Week 12 Follow-up visit to Week 24 Follow-up Visit (approximately 12 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06462700
Number analyzed (Participants) | 3
Participants
  Week 12 Transfusion Independence | 0
  Week 24 Transfusion Independence | 2

ADVERSE EVENTS:
Time Frame: Screening up to 24 weeks of follow-up (approximately up to 28 weeks)
Arm/Group | PF-06462700
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06462700 (N=3)
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Feeling abnormal (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Oedema (General disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Serum sickness (Immune system disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Oxygen saturation abnormal (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT04350606/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT04350606/SAP_001.pdf